CLINICAL TRIAL: NCT06330740
Title: Reducing Medication Ordering Errors Through Indications-Based Prescribing
Brief Title: Evaluations of CDS Systems
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Presbyterian Hospital (Other)
Responsible Party: Principal Investigator, Anne Grauer, Assistant Professor of Clinical Medicine at CUIMC, New York Presbyterian Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAU3416
Record Dates: First submitted 2023-12-28; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Safety Issues
Keywords: medication safety; patient safety

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental)
  Interventions: Other: Clinical Decision Support
- Control Arm (No Intervention)

INTERVENTIONS:
Other: Clinical Decision Support — Upon ordering antibiotics the provider will be prompted to utilize an indication-based order set which guides the clinician to the appropriate empiric antibiotic choice.
  Arms: Intervention Arm

SUMMARY:
Indications-based prescribing is a medication ordering system in which a clinician selects an indication, and then the electronic health record (EHR) suggests an appropriate medication regimen. This approach was shown to significantly decrease medication ordering errors in a prototype environment. However, the effect of indications-based prescribing on preventing ordering errors has not been rigorously evaluated in a real-world healthcare setting. Antibiotics are the medication class most likely to contain ordering errors, which can lead to significant patient harm. At NewYork-Presbyterian (NYP) a robust antimicrobial indication-based order set was developed to help clinicians identify the appropriate antibiotic, dose, frequency, and duration, based on type of infection and patient-specific characteristics, but it is not widely used. The investigators propose a randomized controlled trial to assess the effectiveness of this indications-based order set for reducing antimicrobial ordering errors.

ELIGIBILITY:
Inclusion Criteria:

All providers placing inpatient orders on adult patients.

Exclusion Criteria:

Providers placing orders on patients who were ordered for antibiotics >24 hours in the past 72 hours and/or patients with positive cultures during that admission, and/or placing an order from the order set.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The combined rate of Wrong Drug, Wrong Duration, Wrong Dose and Wrong Frequency Retract-And-Reorder (RAR) events will be combined to create an overall rate of near-miss ordering errors in the control and intervention arm. | Up to 18 months
  Novel Health IT measures which utilize provider ordering patterns to capture near-miss ordering errors.

IPD SHARING:
Plan to Share IPD: No